CLINICAL TRIAL: NCT01454635
Title: Treatment Response Study of Sertraline to Treat Japanese Major Depressive Disorder
Brief Title: Analisis of Facors Involved in Antidepressant Treatment Response of Major Depressive Disorder
Acronym: AFADTRMDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa University (Other)
Responsible Party: Principal Investigator, Gentaro Nishioka, Tokyo Metropolitan Police Hospital, Department of Psychiatry, Principal Investigator, Showa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-GEC-84
Record Dates: First submitted 2011-10-17; First posted 2011-10-19 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Major Depressive Disorder
Keywords: depression; treatment response; selective serotonin reuptake inhibitor
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertraline, Treatment response (Other): dosage, frequency and duration
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — dosage,frequency and duration
  Other Names: J Zoloft®

SUMMARY:
The purpose of this study is to predict and visualize sertraline treatment response in major depressive disorder with clinical symptoms, demographic and stress state, personality, eight genetic polymorphisms at baseline.

DETAILED DESCRIPTION:
While only about 50% of patients respond to first treatment in major depressive disorder, 30-40% did not remit after continuous 1 year treatment. However, patients must remain on their prescribed medications for at least 4 weeks without knowing whether the particular antidepressant will be effective. Studies have suggested a number of predictors of treatment response, but varying degrees of success and nearly all with poor prognostic sensitivity and specificity. The investigators investigated clinical symptoms, demographic and stress state, personality and genetic polymorphisms in patients of major depressive disorder treated with sertraline and performed multivariate analysis to extract the predicting factors. Moreover, the investigators tried to visualize weight of variables and pathway one another.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Major Depressive Disorder
* Must be able to swallow tablets

Exclusion Criteria:

* pregnant
* breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kiuchi, Professor, Study Director — Showa University
Locations (1):
- Showa University Northern Yokohama Hospital, Yokohama, Kanagawa, Japan